CLINICAL TRIAL: NCT05195970
Title: Microbiota, Metabolites and Colon Neoplasia
Brief Title: Walnuts and Colon Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Weill Medical College of Cornell University (Other); University of Connecticut (Other); California Walnut Commission (Other); Spanish National Research Council (Other Government); University of Florida (Other)
Responsible Party: Principal Investigator, Daniel Rosenberg, Professor of Medicine, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-167JS-1; 1R01CA252045-01A1 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2022-01-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Diet Habit
Keywords: Colorectal cancer; Microbiome; Urolithin; Walnuts; Diet habit; Inflammatory markers; Colon inflammation
MeSH Terms: conditions — Colorectal Neoplasms; Feeding Behavior; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Walnut Consumption (Experimental): Following enrollment, participants will start a 7-day wash-out period where they will be asked to avoid foods and beverages high in ellagitannins. These include pomegranates, hazelnuts, pistachios, walnuts (besides the samples given by the researchers), strawberries, raspberries, blackberries, oak-aged wines and spirits; a full list of foods and beverages to avoid will be provided. Then, participants will consume 2 ounces of walnuts daily with their usual diet while continuing to avoid ellagitannins for 21 days prior to their routine colonoscopy.
  Interventions: Other: Walnuts

INTERVENTIONS:
Other: Walnuts — Participants consume 2 ounces of walnuts daily for 21 days

SUMMARY:
The purpose of this research study is to examine whether adding walnuts to your diet can have a beneficial effect on the gut bacteria population, inflammatory markers in the blood, and the tissue that lines the inside of the colon.

DETAILED DESCRIPTION:
This is a 30-day dietary intervention study where participants will be asked to consume 2 ounces of walnuts daily for 21 days, and at the end of the study period they will come in for a routine colonoscopy. After being informed about the study and potential risks, participants giving written informed consent will first start a 7-day wash-out period where they will be asked to avoid foods high in ellagitannins for the duration of the study. In addition, participants will be asked to complete food and activity questionnaires, a walnut consumption log, and two sets of 3-day dietary records during their participation in the study. Participants will also be asked to provide three urine samples, two blood samples, and two stool samples at multiple time points, and 8-10 colon tissue specimens (biopsies) will be collected during their colonoscopy procedure for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 39-75 years old who meet the criteria of one of the following groups and are eligible to undergo a routine screening or surveillance colonoscopy for colorectal cancer (CRC):

   1. Individuals who have a family history of colon polyps or CRC in a first-degree relative diagnosed with CRC under the age of 65 years, or
   2. Individuals who are referred for colonoscopy following a positive fecal immunochemical test (FIT) or a positive Cologuard screening test and have not had a high-quality colonoscopy in the past 3 years, or
   3. Individuals who have a personal history of colon polyps
2. Willing and able to provide written informed consent for study participation
3. Willing to consume 2 ounces (56 grams) of walnuts daily for 3 weeks
4. Willing to avoid intake of EA/ET-rich foods and beverages (e.g., pomegranates, hazelnuts, pistachios, strawberries, raspberries, blackberries, oak-aged wines, and other items on a list given by researchers) and fermented dairy products containing viable Bifidobacteria or Lactobacilli)
5. Willing to stop taking dietary supplements, including probiotics
6. Willing to have two separate blood draws, as well as urine and stool collections
7. Willingness to comply with all study requirements

Exclusion Criteria:

1. Individual has a personal history of CRC, or a history of any malignancy (other than skin cancer) within the past 5 years
2. Individual meets the Amsterdam criteria for Lynch Syndrome or has a history of familial adenomatous polyposis (FAP)
3. Individual has been treated with immunosuppressive agents or systemic steroids, excluding inhalers, at least two weeks prior to the Screening Visit and for the duration of the study
4. Use of antibiotics at least one month prior to the Screening Visit and for the duration of the study
5. Patients with severe medical illness or those at high risk for anesthesia, as determined by good clinical practice
6. Current evidence or previous history of ulcerative colitis or Crohn's disease
7. Colonoscopy performed for reasons other than screening or surveillance for CRC
8. HIV infection, chronic viral hepatitis
9. Allergy to walnuts or hypersensitivity to tree nuts
10. Peri-menopausal women with any chance or plan of pregnancy
11. Individuals with blood coagulation disorders or on anti-coagulant therapy
12. Any other condition that, in the opinion of the PI, might interfere with study objectives
13. No race/ethnicity, language or gender exclusions for this study

Ages: 39 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial composition and taxonomy changes in the fecal microbiome | Day 7 and Day 28
  Bacterial composition and taxonomy changes in the fecal microbiome will be assessed using 16 Svedberg unit (16S) ribosomal ribonucleic acid (rRNA) sequencing, at day 7 (post-washout/pre-walnut supplementation) and at day 28 (post-walnut supplementation).
Bacterial diversity changes and strain-level variations in the fecal microbiome | Day 7 and Day 28
  Bacterial diversity/abundance changes and strain-level variations in the fecal microbiome will be assessed using metagenomic shotgun sequencing at day 7 (post-washout/pre-walnut supplementation) and at day 28 (post-walnut supplementation).
Bacterial gene expression profile changes in the fecal microbiome | Day 7 and Day 28
  Bacterial gene expression profile changes in the fecal microbiome will be assessed using metagenomic ribonucleic acid (RNA) sequencing at day 7 (post-washout/pre-walnut supplementation) and at day 28 (post-walnut supplementation).
Urolithin levels in urine | Day 0, Day 7 and Day 30
  Urolithin levels will be measured in urine by ultra-high performance liquid chromatography with quadrupole time-of-flight mass spectrometry at day 0 (baseline/pre-washout), day 7 (post-washout/pre-walnut supplementation) and day 30 (post-walnut supplementation/end of study).
Association of urolithin levels with presence (and type) of colonic lesions | Day 30
  Baseline urolithin levels measured in the urine by ultra-high performance liquid chromatography with quadrupole time-of-flight mass spectrometry will be associated with the presence (and type) of colonic lesions (e.g., advanced adenomas (AAs) or sessile serrated adenomas/polyps (SSA/Ps)) detected during the colonoscopy procedure at the end of the study (day 30).
Correlation of urolithin levels with fecal microbiome composition | Day 7 and Day 28
  Detailed statistical analyses will be used to correlate urolithin formation with the composition of the fecal microbiome at day 7 (post-washout/pre-walnut supplementation) and at day 28 (post-walnut supplementation).
Correlation of colonic lesion gene expression with urolithin production | Day 30
  Colonic lesion (AAs and SSA/Ps) biopsies obtained at the end of the study (day 30) during the colonoscopy procedure will undergo DNA sequence-based analysis to determine gene expression profiling. These results will be compared to urinary urolithin levels measured at baseline to establish correlations between urolithin production and colorectal cancer risk markers.
Association of urolithin levels with the immune composition of the tumor microenvironment | Day 30
  FFPE colon polyp tissue sections will be analyzed by the NCI Imaging Core (Frederick, MD) using imaging mass cytometry (IMC) to determine immune cell populations present within the tumor microenvironment. This data will be used to establish correlations with urolithin production.

SECONDARY OUTCOMES:
Short-chain fatty acid composition in stool | Day 7 and Day 30
  Short-chain fatty acids in freeze-dried stool samples will be measured using differential mobility separation at day 7 (post-washout/pre-walnut supplementation) and at day 30 (post-walnut supplementation).
Bile acid metabolism in stool | Day 7 and Day 30
  Primary and secondary bile acids in freeze-dried stool samples will be analyzed using standard liquid chromatography-mass spectrometry methods at day 7 (post-washout/pre-walnut supplementation) and at day 30 (post-walnut supplementation).
Inflammatory markers in blood | Day 7 and Day 30
  Markers of systemic inflammation associated with adenoma risk will be measured in plasma using commercial enzyme-linked immunoassay (ELISA) kits at day 7 (post-washout/pre-walnut supplementation) and at day 30 (end of study).
Correlation of dietary behavior with presence (or absence) of colonic polyps | Day 7 and Day 30
  Overall diet quality and habits documented on brief food questionnaires will be analyzed by NutritionQuest at day 7 (post-washout/pre-walnut supplementation). Dietary behavior data will be correlated with the presence or absence of colonic polyps detected during the colonoscopy procedure at the end of the study (day 30).
Correlation of dietary behavior with fecal microbiome composition and diversity | Day 7 and Day 30
  Dietary behavior data documented on 3-day dietary records will be analyzed by Nutrition Data System for Research software. This data will be correlated with fecal microbiome composition and diversity at day 7 (post-washout/pre-walnut supplementation) and at day 30 (post-walnut supplementation).
Correlation of dietary behavior with urolithin production | Day 7 and Day 30
  Dietary behavior data documented on 3-day dietary records will be analyzed by Nutrition Data System for Research software. This data will be correlated with urolithin levels at day 7 (post-washout/pre-walnut supplementation) and at day 30 (post-walnut supplementation).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W. Rosenberg, Ph.D., Principal Investigator — UConn Health; Christian Jobin, Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UConn Health, Farmington, Connecticut
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan N, Fusco JL, Rosenberg DW. Antioxidant and Anti-Inflammatory Properties of Walnut Constituents: Focus on Personalized Cancer Prevention and the Microbiome. Antioxidants (Basel). 2023 Apr 22;12(5):982. doi: 10.3390/antiox12050982. PMID 37237848
- [Background] Liu H, Birk JW, Provatas AA, Vaziri H, Fan N, Rosenberg DW, Gharaibeh RZ, Jobin C. Correlation between intestinal microbiota and urolithin metabolism in a human walnut dietary intervention. BMC Microbiol. 2024 Nov 15;24(1):476. doi: 10.1186/s12866-024-03626-5. PMID 39548408
- [Background] Moussa MR, Fan N, Birk J, Provatas AA, Mehta P, Hatano Y, Chun OK, Darooghegi Mofrad M, Lotfi A, Aksenov A, Motta VN, Zenali M, Vaziri H, Grady JJ, Nakanishi M, Rosenberg DW. Systemic Inflammation and the Inflammatory Context of the Colonic Microenvironment Are Improved by Urolithin A. Cancer Prev Res (Phila). 2025 Apr 1;18(4):235-250. doi: 10.1158/1940-6207.CAPR-24-0383. PMID 39995164
- [Background] Nakanishi M, Matz A, Klemashevich C, Rosenberg DW. Dietary Walnut Supplementation Alters Mucosal Metabolite Profiles During DSS-Induced Colonic Ulceration. Nutrients. 2019 May 20;11(5):1118. doi: 10.3390/nu11051118. PMID 31137456
- [Background] Chen Y, Nakanishi M, Bautista EJ, Qendro V, Sodergren E, Rosenberg DW, Weinstock GM. Colon Cancer Prevention with Walnuts: A Longitudinal Study in Mice from the Perspective of a Gut Enterotype-like Cluster. Cancer Prev Res (Phila). 2020 Jan;13(1):15-24. doi: 10.1158/1940-6207.CAPR-19-0273. Epub 2019 Dec 9. PMID 31818852
- [Background] Nakanishi M, Chen Y, Qendro V, Miyamoto S, Weinstock E, Weinstock GM, Rosenberg DW. Effects of Walnut Consumption on Colon Carcinogenesis and Microbial Community Structure. Cancer Prev Res (Phila). 2016 Aug;9(8):692-703. doi: 10.1158/1940-6207.CAPR-16-0026. Epub 2016 May 23. PMID 27215566
- [Background] Hong BY, Ideta T, Lemos BS, Igarashi Y, Tan Y, DiSiena M, Mo A, Birk JW, Forouhar F, Devers TJ, Weinstock GM, Rosenberg DW. Characterization of Mucosal Dysbiosis of Early Colonic Neoplasia. NPJ Precis Oncol. 2019 Nov 14;3:29. doi: 10.1038/s41698-019-0101-6. eCollection 2019. PMID 31754633
- [Background] Tomas-Barberan FA, Gonzalez-Sarrias A, Garcia-Villalba R, Nunez-Sanchez MA, Selma MV, Garcia-Conesa MT, Espin JC. Urolithins, the rescue of "old" metabolites to understand a "new" concept: Metabotypes as a nexus among phenolic metabolism, microbiota dysbiosis, and host health status. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201500901. Epub 2016 Jun 20. PMID 27158799